CLINICAL TRIAL: NCT03436797
Title: An Open-Label, Pilot Study to Assess the Efficacy and Safety of AK002 (Siglec-8) in Subjects With Antihistamine-Resistant Chronic Urticaria
Brief Title: A Study to Assess the Efficacy and Safety of AK002 in Subjects With Antihistamine-Resistant Chronic Urticaria
Acronym: CURSIG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK002-006
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — AK002

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK002-IV (Experimental): AK002 given as monthly intravenous infusions at up to 3 mg/kg.
  Interventions: Drug: AK002

INTERVENTIONS:
Drug: AK002 — AK002 is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8, a member of the CD33-related family of sialic acid-binding, immunoglobulin-like lectins (Siglecs).

SUMMARY:
This is a Phase 2a, open-label study to assess the effects of AK002

DETAILED DESCRIPTION:
This open-label study is to assess the effects of AK002, given as monthly intravenous infusions at up to 3 mg/kg. A total of 47 patients will be enrolled across 2-4 sites. All patients enrolled in the study will receive 6 monthly infusions of AK002 and will then be followed for another 8 weeks. Some patients will have the option to receive an additional 12 months of extended dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 and ≤ 85 years old)
2. Body weight <125 Kg
3. Informed consent signed and dated
4. Able to read, understand, and willing to sign the informed consent form and comply with study procedures
5. Diagnosis of CU for at least three months, refractory to antihistamine treatment in single or 4-fold dosage
6. Willing, committed, and able to return for all clinic visits and complete all study-related procedures, including willingness to have IV infusion of study drug administered by a qualified person
7. Females of childbearing potential must have a negative pregnancy test at Baseline. Female subjects must be willing to use highly effective contraception (Pearl- 4 Index < 1). A woman will be considered not of childbearing potential if she is post-menopausal for greater than two years (FSH >40mL) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)
8. No participation in other clinical trials 4 weeks before participation in this study
9. Uncontrolled CU (UCT <12) at the time of enrollment

Exclusion Criteria:

1. Acute urticaria
2. Concurrent/ongoing treatment with immunosuppressives (e.g., cyclosporine, methotrexate, dapsone, or others) within 4 weeks or 5 half-lives prior to Baseline, whichever is longer
3. Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial
4. Significant concomitant illness that would adversely affect the subject's participation or evaluation in this study
5. History of malignancies within five years prior to screening other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cancer
6. Presence of clinically significant laboratory abnormalities
7. Lactating women or pregnant women
8. Substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) within the last 5 years that could limit the subject's ability to comply with study procedures
9. Subjects who are detained officially or legally to an official institute or those that have been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities will be excluded from the study
10. Use of omalizumab within the last 3 months
11. Receipt of intravenous IgG therapy 30 days prior to Baseline
12. Plasmapheresis 30 days prior to Baseline
13. Use (daily or every other day) of Doxepin 14 days prior to Baseline
14. Receipt of inactive vaccination or live attenuated vaccine 30 days prior to Baseline
15. Use of H2 antihistamines 7 days before Baseline
16. Intake of leukotriene antagonists within 7 days prior to enrollment
17. Intake of systemic corticosteroids (e.g., oral or depot) within 14 days prior to enrollment
18. Positive screening for ova and parasite test at Baseline
19. Treatment of helminthic parasite within 6 months of screening
20. Positive HIV serology at screening
21. Positive Hepatitis serology at baseline, except for vaccinated patients or patients with past but resolved hepatitis at screening
22. Donation or loss of >500ml of blood within 56 days prior to administration of study drug or donation of plasma within 7 days prior to administration of drug
23. Known hypersensitivity to any ingredients of AK002 or drugs related to AK002 (e.g., monoclonal antibodies, polyclonal gamma globulin)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Director — Allakos Inc.
Locations (4):
- United States (2):
  - Allakos Investigational Site, Edgewater, Florida
  - Allakos Investigational Site, Cincinnati, Ohio
- Germany (2):
  - Allakos Investigational Site, Berlin
  - Allakos Investigational Site, Mainz

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 subjects were enrolled in the main study and received at least one dose of AK002. 45 subjects had at least one post-baseline assessment of the primary efficacy variable and were reported in the baseline period. 5 subjects from the main study were allowed the option to receive extended dosing with up to 12 additional doses of AK002.
Pre-assignment Details: no pre-assignment was done
Groups:
- AK002: For the main study phase, single doses of AK002 were administered by IV infusion every 28 days at Weeks 0, 4, 8, 12, 16, and 20. For the extended dosing phase, single doses of AK002 were administered by IV infusion on Extended Dosing Days 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, and 309.
  The arm included all subjects who were enrolled.
Period: Main Study
Arm/Group | AK002
Started | 47 (47 subjects were enrolled in this study and received at least one dose of the study drug. 45 of these subjects had at least one post-baseline assessment of the primary efficacy variable and were reported in the baseline period.)
Completed | 37
Not Completed | 10
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Non-Specific | 2
Period: Extended Dosing
Arm/Group | AK002
Started | 5 (5 subjects in the CholU, UF, and CSU-XOLAIR® (omalizumab) failure cohorts of the main study who received all 6 infusions of AK002, were followed at least through Day 155, and demonstrated severe symptoms of urticaria following the last dose of treatment were allowed the option to receive extended dosing with up to 12 additional doses of AK002.)
Completed | 4
Not Completed | 1
Not completed — Patient decision | 1

BASELINE CHARACTERISTICS:
Population: 47 subjects were enrolled in the main study and received at least one dose of the study drug; 45 of these subjects had at least one post-baseline assessment of the primary efficacy variable and were reported in the baseline period. 5 subjects in the CholU, UF, and CSU-XOLAIR® (omalizumab) failure cohorts of the main study were enrolled in the extended dosing phase.
Groups:
- AK002: For the main study, single doses of AK002 were administered by IV infusion every 28 days at Weeks 0, 4, 8, 12, 16, and 20. The arm included all subjects who were enrolled in the main study, did receive at least 1 dose of the study drug, and had at least 1 post-baseline assessment of the primary efficacy variable (=modified intention-to-treat population, mITT).
  For the extended dosing phase, the arm included all subjects who were enrolled in the extended dosing and received at least 1 dose of the study drug.
Arm/Group | AK002
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] — Population: 45 subjects in the Main Study Phase. 5 subjects entered the Extended Dosing Phase.
  years
    Main Study Phase | 42 [18 to 75]
    Extended Dosing Phase: number analyzed (Participants) | 5
    Extended Dosing Phase | 43 [24 to 55]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 45 subjects in the Main Study Phase. 5 subjects entered the Extended Dosing Phase.
  Participants
    Main Study Phase: Female | 34
    Main Study Phase: Male | 11
    Extended Dosing Phase: number analyzed (Participants) | 5
    Extended Dosing Phase: Female | 5
    Extended Dosing Phase: Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 45 subjects in the Main Study Phase. 5 subjects entered the Extended Dosing Phase.
  Participants
    Main Study Phase: Hispanic or Latino | 2
    Main Study Phase: Not Hispanic or Latino | 43
    Main Study Phase: Unknown or Not Reported | 0
    Extended Dosing Phase: number analyzed (Participants) | 5
    Extended Dosing Phase: Hispanic or Latino | 1
    Extended Dosing Phase: Not Hispanic or Latino | 4
    Extended Dosing Phase: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 45 subjects in the Main Study Phase. 5 subjects entered the Extended Dosing Phase.
  Participants
    Main Study Phase: American Indian or Alaska Native | 0
    Main Study Phase: Asian | 0
    Main Study Phase: Native Hawaiian or Other Pacific Islander | 0
    Main Study Phase: Black or African American | 1
    Main Study Phase: White | 44
    Main Study Phase: More than one race | 0
    Main Study Phase: Unknown or Not Reported | 0
    Extended Dosing Phase: number analyzed (Participants) | 5
    Extended Dosing Phase: American Indian or Alaska Native | 0
    Extended Dosing Phase: Asian | 0
    Extended Dosing Phase: Native Hawaiian or Other Pacific Islander | 0
    Extended Dosing Phase: Black or African American | 0
    Extended Dosing Phase: White | 5
    Extended Dosing Phase: More than one race | 0
    Extended Dosing Phase: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — This is the region of enrollment for the Main Study Phase. In the Extended Dosing Phase, all 5 subjects were from Germany.
  Participants
    United States | 16
    Germany | 29
Urticaria Control Test (UCT) Score [Mean (Standard Deviation); unit: Score on a scale] — Population: 45 subjects in the Main Study Phase. 5 subjects entered the Extended Dosing Phase.
  Score on a scale
    Main Study Phase | 4.4 (3.1)
    Extended Dosing Phase: number analyzed (Participants) | 5
    Extended Dosing Phase | 1.6 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Urticaria Control Test (UCT) Score From Baseline to Week 22 in the Main Study Phase
Description: The UCT score consists of 4 items, and each UCT item has 5 answer options (scored with 0-4 points), where low points indicate high disease activity and low disease control of chronic urticaria. The UCT score, ranging from 0 to 16, is calculated by adding all 4 individual item scores. A UCT score of 16 points indicates complete disease control and a change of the UCT score of 3 or more points was regarded as clinically relevant (minimal clinically important difference [MCID]).
Time Frame: Baseline to Week 22 (Main Study Phase)
Population: Modified intention-to-treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- CholU: The CholU cohort included subjects with Cholinergic Urticaria.
- UF-Cohort: The UF cohort included subjects with Urticaria Factitia.
- CSU-XN: The CSU-XN cohort included XOLAIR® (omalizumab) naïve subjects with Chronic Spontaneous Urticaria (CSU).
- CSU-XF: The CSU-XF cohort included subjects with Chronic Spontaneous Urticaria (CSU) who did not achieve an adequate response to XOLAIR® (omalizumab) in the opinion of the Investigator.
Arm/Group | CholU | UF-Cohort | CSU-XN | CSU-XF
Number analyzed (Participants) | 11 | 10 | 13 | 11
Score on a scale | 6.5 (6.15) | 3.4 (4.09) | 11.1 (4.07) | 4.8 (6.97)

2. Other Pre Specified Outcome: Safety and Tolerability of up to 12 Additional Doses of AK002 in Subjects With CU in the Extended Dosing Phase
Description: Adverse events were assessed during the Extended Dosing Phase of the study, and only the 5 subjects who entered the Extended Dosing Phase were included.
Time Frame: Through study completion, up to 52 weeks (Extension Dosing Phase)
Population: 5 subjects from the main study were enrolled in the Extended Dosing Phase.
Measure: Count of Participants; unit: Participants
Groups:
- AK002: The arm included all subjects who were enrolled in the Extended Dosing Phase.
Arm/Group | AK002
Number analyzed (Participants) | 5
Participants
  Subjects with ≥1 adverse events | 5
  Subjects with ≥1 treatment-related adverse events | 4
  Subjects with an adverse event leading to study drug discontinuation | 0
  Subjects with ≥1 serious adverse events | 1
  Subjects with ≥1 treatment-related serious adverse events | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the first dose of AK002 until the end of Follow-up (Week 28 in the Main Study Phase, Week 52 in the Extended Dosing Phase).
Description: Adverse events were reported systematically.
Groups:
- AK002 Main Study: This arm included all subjects who were enrolled in the Main Study Phase
- AK002 Extended Dosing: This arm included all subjects from the main study who were enrolled in the Extended Dosing Phase
Arm/Group | AK002 Main Study | AK002 Extended Dosing
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/47 | 1/5
Other Adverse Events (participants affected / at risk) | 33/47 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AK002 Main Study (N=47) | AK002 Extended Dosing (N=5)
Hypertension (Vascular disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AK002 Main Study (N=47) | AK002 Extended Dosing (N=5)
Chest pain (General disorders) | 3 | 0
Fatigue (General disorders) | 3 | 0
Influenza like illness (General disorders) | 3 | 0
Pyrexia (General disorders) | 3 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 20 | 3
Headache (Nervous system disorders) | 9 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Nasopharyngitis (Infections and infestations) | 10 | 4
Sinusitis (Infections and infestations) | 3 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 1
Goitre (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Inflammation (General disorders) | 1 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 0 | 2
Tinea manuum (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (2):
  • Study Protocol (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT03436797/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03436797/SAP_001.pdf